CLINICAL TRIAL: NCT07081789
Title: The Effect of Listening to Music and Making Puzzles in Cope With Dysmenorrhea in Young Women: A Randomized Controlled Study
Brief Title: Music and Puzzle Use in Dysmenorrhea Relief
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Burdur Mehmet Akif Ersoy University (Other)
Responsible Party: Principal Investigator, ENDAM ÇETİNKAYA AK, Assistant Professor, Burdur Mehmet Akif Ersoy University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: GO 2024/843
Record Dates: First submitted 2025-06-30; First posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Dysmenorrhea
Keywords: Dysmenorrhea; Pain; Puzzle; Music; Complementary medicine
MeSH Terms: conditions — Dysmenorrhea; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Music Group (Experimental)
  Interventions: Behavioral: Music Listening
- Puzzle Group (Experimental)
  Interventions: Behavioral: Puzzle Activity
- Control Group (No Intervention): No intervention.

INTERVENTIONS:
Behavioral: Music Listening — Participants will listen to a 24 min 54 sec music track for 4 days (starting 3 days before menstruation).
  Arms: Music Group
Behavioral: Puzzle Activity — Participants will do puzzles for the same duration and timing.
  Arms: Puzzle Group

SUMMARY:
The aim of this clinical trial is to evaluate whether interventions such as listening to music and doing puzzles are effective in reducing menstrual pain, menstrual symptoms, and perceived stress in young women with dysmenorrhea, ages 18-25.

The main questions it aims to answer are:

Do listening to music and doing puzzles reduce dysmenorrhea pain? Do these interventions affect menstrual symptoms and perceived stress? The researchers will compare music, puzzle, and control groups to assess the effects on pain intensity, menstrual symptoms, and perceived stress levels.

Participants:

Participants will be followed for three menstrual cycles, In the first cycle, pain, symptoms, and stress levels will be measured,

In the next two cycles:

Music group: Listen to a specific song with headphones for four days, Puzzle group: Do puzzles for the same amount of time, Control group: Measurements only, without intervention.

DETAILED DESCRIPTION:
Objective:This study aimed to determine the effects of listening to music and doing puzzles on coping with dysmenorrhea in young women.

Method The study is a single-center, double-blind, prospective, three-parallel-group randomized controlled trial conducted at a university health school. Participants will be followed for three menstrual cycles. In the first menstrual cycle, menstrual pain, menstrual symptoms, and perceived stress level scales will be administered. In the second and third menstrual cycles, two interventions, doing puzzles and listening to music, will be administered.

A randomization method will be used to assign participants to music, puzzles, or control groups, ensuring that extraneous variables are equally distributed. Blinding procedures will be applied for both participants and researchers to control for bias and confounding factors. Intervention protocols will be standardized to ensure consistency. Inclusion and exclusion criteria were carefully defined to control for variables that could affect the validity of the study.

Universe and Sample/Study Group (The path to be followed in creating the sample and study group should be explained.) The universe of the study will consist of all female students studying at a university's health school, meeting the criteria for inclusion in the study, and agreeing to participate in the study.

The study sample will consist of female students who meet the criteria for inclusion in the study and agree to participate in the study between the dates of the study. The sample size will be calculated by performing a power analysis with the G power program and by taking a study as a reference. It was determined that 28 people from each group would be sufficient to participate in the study with an effect size of 0.75, α = 0.05 margin of error, and minimum power = 80% (β = 0.2%). However, considering possible missing data, it was decided to include 32 female students in the study with a 10% increase in each group.

The simple random sampling method will be used in this study. The study aims will be explained to the female students who are eligible to participate and agree to participate, and they will be informed that they will be randomly assigned to the control group, puzzle group, and music group. However, the study hypothesis will not be disclosed to avoid the expectation bias effect. The study will be conducted with 96 female students with dysmenorrhea, considering the expected 10% loss rate. For randomization; a list of students who meet the study criteria will be created and the students will be divided into three groups from this list using the simple random sampling method. Inclusion Criteria for the Study: Female students studying at a university health school, between the ages of 18-25, with a Visual Analog Scale (100 mmVAS pain) intensity of 5 or above, and with regular menstrual cycles (28 ± 7 days) in the last year will be included in the study. Individuals who do not have pelvic pathology, hearing loss, endocrine, neurological or chronic diseases such as diabetes and heart disease, psychiatric diseases, do not use oral contraceptives or antidepressants, do not have menstrual irregularities, do not have mental problems that prevent evaluation and cooperation, have not undergone pelvic surgery, do not have malignant diseases, do not have obesity, do not have previous pregnancies, do not have advanced musical education, and do not use vitamin supplements will be included.

Participants who do not meet the inclusion criteria, who use medication, nonpharmacological applications (acupressure, reiki, reflexology, meditation) or any nutritional supplements to reduce pain will be excluded from the study. Female students participating in the study will be told that they should not use analgesics in order to evaluate the effectiveness of the applications applied during the study, and that they can use analgesics only if their severe and unbearable pain continues in the pain assessment made after the applications.

A double-blind randomized controlled design will be used in this study. The researchers will contact the students with dysmenorrhea included in the study during the initial data collection phase and during the follow-up of interim measurements. Due to the nature of the double-blind study, the assignment of participants to groups, the implementation of interventions, and the statistical analysis of the research findings will be performed by scientists not involved in the study.

Data Collection Tool The data collection form consists of four sections. The first section consists of the Individual Identification Form, which consists of a total of 28 questions that examine socio-demographic and menstrual cycle-related characteristics and was created by the researchers by reviewing the literature.

The Visual Analog Scale (100 mm VAS pain) is the second part of the questionnaire. The level and severity of menstrual pain will be measured using the 100 mm VAS pain, which is a valid and reliable tool for measuring experimental and clinical pain. The 100 mm VAS pain is scored on a 10 cm horizontal line (0 = no pain and 10 = worst possible pain). In the third part, the Menstrual Symptom Scale (MSS) will be used to assess menstrual symptoms. This scale was developed in English in 1975 to assess menstrual pain and symptoms. It is a widely used scale in the USA and many other countries. In 2009, its factor structure and usability in adolescents were re-evaluated and updated. The scale was adapted to Turkish in 2014. Participants are asked to assign a number between 1 (never) and 5 (always) to the symptoms they experience related to menstruation. Scale items are numbered according to the separated factors for ease of use. Items numbered 1-13 belong to the "Negative effects/somatic complaints" subscale, items numbered 14-19 belong to the "Menstrual pain symptoms" subscale, and items numbered 20-22 belong to the "Coping methods" subscale. It is a five-point Likert-type scale consisting of a total of 22 items. Participants are asked to give a number between 1 (never) and 5 (always) to the symptoms they experience related to menstruation. The score obtained from the sub-dimensions is calculated by taking the average of the total scores of the items in the sub-dimensions. An increase in the average score indicates an increase in the severity of menstrual symptoms. An increase in the average score of the sub-scales indicates an increase in the severity of menstrual symptoms related to that sub-scale. The Cronbach Alpha value of the scale is 0.92. In the fourth section, the Perceived Stress Scale (PSS) will be used to assess the level of perceived stress. The total score that can be obtained from the scale is 32. The scale consists of 10 items and is scored between 0 and 4. A high total score indicates a high stress level. In this study, the scale whose Turkish validity and reliability study was conducted in 2009 was used. The Cronbach alpha value of the scale is 0.86.

Data Collection In the first month of participation in the study, all participants will be assessed for their current pain status, menstrual symptoms, and perceived stress levels before the interventions. In the second and third months, 100 mm VAS pain will be determined on the first day of the menstrual cycle to assess menstrual pain intensity, MBS will be used to assess menstrual symptom status, and PSS will be used to assess perceived stress. When the literature is reviewed, it has been reported that prostaglandin levels are high on the first day of the menstrual cycle, and accordingly, it was considered appropriate to assess the pain of students with dysmenorrhea on the first day of the menstrual cycle.

In order to standardize the evaluation processes of the interventions (music and puzzles) applied to the groups, participants will be asked to do a puzzle and listen to music until noon (12:00) at the latest. Participants in the music and puzzle groups will be asked to evaluate their pain, menstrual symptoms, and perceived stress in the afternoon (after 12:00) following the intervention, and the control group will be asked to evaluate their pain, menstrual symptoms, and perceived stress on the first day when they are most intense. All data will be collected by a researcher.

Music Group In the second and third months when the effectiveness of the study is evaluated, female students will be asked to listen to a song that lasts 24 minutes and 54 seconds, which has been used in studies with high levels of evidence in the literature, for a total of four days, three days before menstruation and the first day of menstruation, using headphones. An anonymous song determined by the researchers after reviewing the literature will be used in the study. The link to access the song will be sent to the participants via social media (WhatsApp). After listening to the music for three days before the menstrual cycle and the first day of menstruation (a total of four days), pain, menstrual symptoms and perceived stress levels on the first day of menstruation will be measured.

Puzzle Group In the second and third months, participants will be asked to do puzzles for 24 minutes and 54 seconds for four days (three days before menstruation and the first day of menstruation) (the duration of the intervention was determined in parallel with the music group so that there was no variability between the groups). The puzzle to be used will be left to the participants' discretion. After doing puzzles three days before the menstrual cycle and the first day of menstruation (a total of four days), pain, menstrual symptoms and perceived stress levels on the first day of menstruation will be measured.

Control group Participants will have their pain, menstrual symptoms and perceived stress levels measured on the first day of their menstrual cycle in the second and third months.

ELIGIBILITY:
Inclusion Criteria

* Female students studying at a university health college
* Female students between the ages of 18 and 25
* Female students with a Visual Analog Scale (100 mmVAS) pain intensity of 5 or higher
* Female students with regular menstrual cycles (28 ± 7 days) within the past year
* Female students without endocrine, neurological, or chronic diseases such as pelvic pathology, hearing loss, diabetes, and heart disease
* Female students without psychiatric illnesses or mental health problems that would interfere with evaluation and cooperation
* Female students who are not using oral contraceptives or antidepressants
* Female students who have not had pelvic surgery
* Female students who have not had malignant diseases
* Female students who are not obese
* Female students who have not previously been pregnant
* Female students who have not received advanced musical training
* Female students who are not taking vitamin supplements

Exclusion Criteria

* Female students who do not meet the inclusion criteria
* Female students who use medication, non-drug practices (acupressure, Reiki, reflexology, meditation), or any nutritional supplements to reduce pain

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Menstrual Pain Severity | Through study completion, an average of 3 mounts
  Menstrual pain intensity will be assessed using the 100 mm Visual Analog Scale (VAS). Participants will rate their pain by marking a point on a 10 cm horizontal line ranging from 0 ("no pain") to 10 ("worst imaginable pain"). Higher scores indicate more severe pain.

SECONDARY OUTCOMES:
Menstrual Symptom Severity | Through study completion, an average of 3 mounts
  Menstrual symptoms will be assessed using the Menstrual Symptom Scale (Menstruasyon Belirti Ölçeği - MBÖ), a 22-item Likert-type questionnaire. Scores range from 1 (never) to 5 (always). Higher total and subscale scores indicate more severe symptoms.
Perceived Stress Level | Through study completion, an average of 3 mounts
  Stress levels will be measured using the 10-item Perceived Stress Scale (PSS). Each item is scored from 0 (never) to 4 (very often), with a total score ranging from 0 to 40. Higher scores indicate higher perceived stress.

CONTACTS AND LOCATIONS:
Overall Officials: Endam Çetinkaya Ak, Assistant Professor, Principal Investigator — Burdur Mehmet Akif Ersoy University
Locations (1):
- Bucak Health School, Burdur, Bucak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data (IPD) will not be shared due to ethical considerations and privacy concerns. The dataset includes sensitive health information, and no data sharing agreements are in place to ensure appropriate secondary use.

REFERENCES:
- [Background] Martin-Saavedra JS, Ruiz-Sternberg AM. The effects of music listening on the management of pain in primary dysmenorrhea: a randomized controlled clinical trial. Nordic J Music Therapy. 2020;29(5):398-415. https://doi.org/10.1080/08098131.2020.1761867.
- [Background] Selçuk AK, Baysal E. The effect of dark chocolate and music on pain and anxiety in young women with primary dysmenorrhea: Randomized controlled trial. Eur J Integr Med. 2022;56:102192. https://doi.org/10.1016/j.eujim.2022.102192.
- [Background] Ferries-Rowe E, Corey E, Archer JS. Primary Dysmenorrhea: Diagnosis and Therapy. Obstet Gynecol. 2020 Nov;136(5):1047-1058. doi: 10.1097/AOG.0000000000004096. PMID 33030880
- [Background] Hu Z, Tang L, Chen L, Kaminga AC, Xu H. Prevalence and Risk Factors Associated with Primary Dysmenorrhea among Chinese Female University Students: A Cross-sectional Study. J Pediatr Adolesc Gynecol. 2020 Feb;33(1):15-22. doi: 10.1016/j.jpag.2019.09.004. Epub 2019 Sep 17. PMID 31539615